CLINICAL TRIAL: NCT06302855
Title: Exploring Adherence and Knowledge Among Diabetic Individuals in Periodontal Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karim Gariani (Other)
Responsible Party: Sponsor-Investigator, Karim Gariani, MD/PhD Head of Diabetes Unit Geneva University Hospital Switzerland, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-00124
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dental visit invited (Active Comparator): Patients will only be invited or asked to schedule a complimentary periodontal check-up visit without any previous assessment.
  Interventions: Diagnostic Test: dental expertise
- dental visit recommended based on dental expertise (Experimental): Patients' oral cavities will be photographed. Based on the remote assessment of periodontitis risk conducted by the same periodontist from the Division of Regenerative Dental Medicine and Periodontology at the University Clinic of Dental Medicine, patients will be invited or asked to schedule a complimentary periodontal check-up visit at the CUMD. The appointment will be arranged directly at the diabetologist's office.
  Interventions: Diagnostic Test: dental expertise

INTERVENTIONS:
Diagnostic Test: dental expertise — dental visit based on dental expertise

SUMMARY:
Objective(s) The primary objective is to evaluate the adherence of diabetic patients to periodontal care, accomplished either through oral communication (group A, control) or through a photograph of their smile, and focusing on their gum health evaluated by a periodontist (group B, test).

Secondary objectives include assessing the prevalence of periodontal disease (PD) in this diabetic sample population and evaluating the presence of specific biomarkers related to it.

The final objective is to assess the agreement between the diagnosis of periodontitis based on the photographs and the diagnosis given after the dental visit, based on the clinical examination. The aim is to determine if the photos could potentially serve as a reliable indicator for periodontal risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes

Exclusion Criteria:

* last dental visit<1 year
* patient unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
adherence of diabetic patients to periodontal | 1 month
  The primary endpoint is to evaluate the adherence of diabetic patients to periodontal care either by informing them orally or after evaluation of their gum health by a periodontist based on a simple photo of their smile.
  .

SECONDARY OUTCOMES:
calculate the prevalence of periodontitis | 1 month
  Secondary endpoints are to calculate the prevalence of periodontitis and the accordance in diagnosis between the photo and the clinical examination of the patient.